CLINICAL TRIAL: NCT03744637
Title: A Study to Assess the Effect of Single Doses of MK-5475 on Pulmonary Vascular Resistance in Patients With Moderate to Severe Pulmonary Arterial Hypertension
Brief Title: A Study of Single Doses of Frespaciguat (MK-5475) on Pulmonary Vascular Resistance (MK-5475-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 5475-002; MK-5475-002 (Other: Merck Study Number)
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Part 1 of the study will evaluate safety, tolerability, and pharmacokinetics in this population using a sequential study design. Review of available safety data up to 24 hours post dose of at least the first 4 participants must occur prior to escalating to the next dose level. A break to review PK data from Periods 1 and 2 will occur after completion of Period 2. Review of safety will occur after completion of Period 3 in all participants from Panel A, prior to initiation of Part 2. An optional break to review rolling PK data from Panel A Period 3 will be dependent upon exposures observed in Periods 1 and 2.
Who Masked: Participant, Investigator
Masking Description: In Part 1 (Panel A) of this study, a double-blinding technique will be used. Frespaciguat and placebo will be packaged identically so that blind is maintained. The participant, the investigator, and Sponsor personnel or delegate(s) who are involved in the study intervention administration or clinical evaluation of the participants are unaware of the intervention assignments.
  Part 2 of this study is conducted as open label; therefore, the Sponsor, investigator, and participant will know the intervention administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Panel A: Frespaciguat 120 ug/165 ug/240 ug/240 ug/240 ug (Parts 1 and 2) (Experimental): Participants in Panel A will receive a single inhaled dose of frespaciguat 120 ug in Period 1 of Part 1, followed by frespaciguat 165 ug in Period 2, followed by frespaciguat 240 ug in Period 3. Each dose will be separated by at least a 7-day washout. In Part 2 Period 2, participants will receive a single inhaled dose of frespaciguat 240 ug and undergo a right heart catheterization (RHC). In Part 2 Period 3, participants will receive a single inhaled dose of frespaciguat 240 ug and undergo a functional respiratory imaging (FRI).
  Interventions: Drug: Frespaciguat
- Panel B: 300 ug/360 ug/360 ug (Part 2) (Experimental): Participants in Panel B will receive a single inhaled dose of frespaciguat 300 ug in Period 1 of Part 2. In Period 2 of Part 2, participants will receive a single inhaled dose of frespaciguat 360 ug and undergo FRI. In Period 3 of Part 2, participants receive a single inhaled dose of frespaciguat 360 ug and undergo RHC. Each dose will be separated by at least a 7-day washout.
  Interventions: Drug: Frespaciguat
- Panel C: 300 ug/360 ug/360 ug (Part 2, Expansion) (Experimental): Participants in Panel C will receive a single inhaled dose of frespaciguat 300 ug in Period 1 of Part 2. In Period 2 of Part 2, participants will receive a single inhaled dose of frespaciguat 360 ug and undergo FRI. In Period 3 of Part 2, participants receive a single inhaled dose of frespaciguat 360 ug and undergo RHC. Each dose will be separated by at least a 7-day washout.
  Interventions: Drug: Frespaciguat
- Panel D: 480 ug/120 ug/120 ug (Part 2) (Experimental): Participants in Panel D will receive a single inhaled dose of frespaciguat 480 ug in Period 1 of Part 2. In Period 2 of Part 2, participants will receive a single inhaled dose of frespaciguat 120 ug and undergo FRI. In Period 3 of Part 2, participants receive a single inhaled dose of frespaciguat 120 ug and undergo RHC. Each dose will be separated by at least a 7-day washout.
  Interventions: Drug: Frespaciguat
- Placebo (Part 1) (Placebo Comparator): Participants will receive a single inhaled dose of matching placebo in Part 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Frespaciguat — Single inhaled dose of frespaciguat 120, 165, 240, 300, 360, or 480 ug depending upon randomization
  Other Names: MK-5475
  Arms: Panel A: Frespaciguat 120 ug/165 ug/240 ug/240 ug/240 ug (Parts 1 and 2); Panel B: 300 ug/360 ug/360 ug (Part 2); Panel C: 300 ug/360 ug/360 ug (Part 2, Expansion); Panel D: 480 ug/120 ug/120 ug (Part 2)
Drug: Placebo — Single inhaled dose of placebo to match frespaciguat
  Arms: Placebo (Part 1)

SUMMARY:
This study of frespaciguat in participants with Group 1 pulmonary arterial hypertension (PAH) will assess the safety, tolerability and pharmacokinetics (PK) of inhaled frespaciguat. There is no formal hypothesis to be tested.

DETAILED DESCRIPTION:
In Part 1, one panel (Panel A) of up to 8 participants will dose in up to 3 dosing periods, with a minimum washout of 7 days between dosing periods. In each dosing period, 6 participants will receive frespaciguat and 2 will receive placebo, with 2 different participants receiving placebo in each of the dosing periods. Review of available safety data will occur prior to escalating to the next dose level.

Participants from Part 1 may continue into Part 2, which will assess safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single-dose inhaled frespaciguat. Three additional panels of participants (Panels B, C and D) will be enrolled into Part 2. Participants in Panel A will participate in 2 open-label dosing periods to assess PD measures associated with right heart catherization (RHC) [Period 2] and functional respiratory imaging (FRI) [Period 3]. Participants in Panels B, C, and D will participate in 3 dosing periods: Period 1 (open-label assessment of safety/tolerability and PK), Period 2 (FRI period) and Period 3 (RHC period).

ELIGIBILITY:
Inclusion Criteria:

* Be or have suspected Group 1 pulmonary hypertension as defined by the Nice 2013 Clinical Classification, including: idiopathic PAH, heritable PAH, drug- or toxin-induced PAH, or PAH associated with connective tissue disease or congenital heart disease
* Have a Body Mass Index (BMI) ≤35 kg/m2,
* Female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: She is a woman of nonchildbearing potential (WONCBP) or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis)
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 14 days, corresponding to time needed to eliminate study intervention(s) after the last dose of study intervention: Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use contraception unless confirmed to be azoospermic (Vasectomized) or secondary to medical cause.
* Have a clinical indication for right heart catheterization (RHC) as part of initial work-up or ongoing medical management
* Panel A: Have history of RHC within 3 years of starting study medication demonstrating mean pulmonary artery pressure of ≥ 27 mmHg and pulmonary vascular resistance (PVR) of ≥ 300 dynes/sec/cm5
* Panels B/C/D: Have history of RHC within 3 years of starting study medication demonstrating mean pulmonary artery pressure of ≥ 27 mmHg and PVR of ≥ 300 dynes/sec/cm5 OR have an echocardiogram performed by the investigator at screening or within 1 year of screening demonstrating pulmonary artery systolic pressure ≥ 50 mmHg in conjunction with 1 or more of the following: tricuspid regurgitation velocity > 3.0 m/s and or significant right heart enlargement and or reduced right heart function.

Exclusion Criteria:

* Has pulmonary hypertension subtypes including the following according to Nice 2013 Clinical Classification: human immunodeficiency (HIV) infection, portal hypertension, schistosomiasis, chronic hemolytic anemia, pulmonary veno-occlusive disease (PVOD) and or pulmonary capillary hemangiomatosis (PCH), persistent pulmonary hypertension of the newborn (PPHN), pulmonary hypertension owing to left heart diseases, left ventricular systolic dysfunction, left ventricular diastolic dysfunction, valvular disease, congenital/acquired left heart inflow/outflow tract obstruction and congenital cardiomyopathies, pulmonary hypertension owing to lung diseases and/or hypoxia, Chronic obstructive pulmonary disease, Interstitial lung disease, other pulmonary diseases with mixed restrictive and obstructive pattern, sleep-disordered breathing, alveolar hypoventilation disorders, chronic exposure to high altitude, developmental abnormalities, pulmonary hypertension defined as chronic thromboembolic pulmonary hypertension [CTEPH]), pulmonary hypertension with unclear multifactorial mechanisms, hematologic disorders: chronic hemolytic anemia, myeloproliferative disorders, splenectomy, systemic disorders: sarcoidosis, pulmonary Langerhans cell histiocytosis, lymphangioleiomyomatosis, neurofibromatosis, vasculitis, metabolic disorders: glycogen storage disease, Gaucher disease, thyroid disorders, others: tumoral obstruction, fibrosing mediastinitis, chronic renal failure, segmental pulmonary hypertension
* Has a history of clinically significant endocrine (not including stable diabetes mellitus), gastrointestinal, cardiovascular, hematological, hepatic (not including chronic stable Hepatitis B and Hepatitis C), immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated, has significant emotional problems
* History of cancer (malignancy) except nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies which have been successfully treated 10 years prior to screening
* History of significant multiple and/or severe allergies
* Known hypersensitivity to iodine or iodine containing products
* Positive for HIV
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks of screening
* Has persistent or permanent atrial fibrillation with an uncontrolled ventricular rate
* Has significantly impaired gas exchange
* Has an active respiratory infection (e.g. common cold, bronchitis, influenza, pneumonia) with lung function outside of the normal range
* Is currently on monotherapy calcium channel blockers as a specific treatment for pulmonary hypertension
* Has taken nitrates within 24 hours of anticipated dosing
* Has taken inhaled prostacyclin within 24 hours of anticipated dosing (iloprost or treprostinil)
* Has taken diltiazem immediate release taken within 24 hours or extended release taken within 48 hours of anticipated dosing
* Has taken sildenafil or vardenafil within 24 hours or tadalafil within 7 days of anticipated dosing
* Has taken soluble guanylate cyclase (sGC) activator for PAH within 24 hours of anticipated dosing
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatment periods), until the poststudy visit
* Has participated in another investigational study within 4 weeks
* Does not agree to follow the smoking restrictions
* Part 2 only: Suffers from claustrophobia and would be unable to undergo computerized tomography (CT) scan
* Part 2 only: Has participated in a positron-emission tomography (PET) research study or other study involving administration of a radioactive substance or ionizing radiation within 12 months prior to the screening visit, or has undergone or plans to have extensive radiological examination within this period
* Consumes greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 12 months. Participants must have a negative urine drug screen (UDS) prior to randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Republican Clinical Hospital of Moldova ( Site 0001), Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Bajwa EK, Cislak D, Palcza J, Feng HP, Messina EJ, Reynders T, Denef JF, Corcea V, Lai E, Stoch SA. Effects of an inhaled soluble guanylate cyclase (sGC) stimulator MK-5475 in pulmonary arterial hypertension (PAH). Respir Med. 2023 Jan;206:107065. doi: 10.1016/j.rmed.2022.107065. Epub 2022 Nov 29. PMID 36521262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with Group 1 Pulmonary Arterial Hypertension (PAH) were recruited to evaluate safety, pharmacokinetics (PK), Functional Respiratory Imaging (FRI), and Right Heart Catheterization (RHC) of single-dose MK-5475.
Groups:
- MK-5475 120 ug/MK-5475 165 ug/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A): Participants received inhaled doses as follows: MK-5475 120 ug (Part 1 Period 1), MK-5475 165 ug (Part 1 Period 2), MK-5475 240 ug (Part 1 Period 3), MK-5475 240 ug (Part 2 Period 2), and MK-5475 240 ug (Part 2 Period 3).
- MK-5475 120 ug/Placebo/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A): Participants received inhaled doses as follows: MK-5475 120 ug (Part 1 Period 1), placebo (Part 1 Period 2), MK-5475 240 ug (Part 1 Period 3), MK-5475 240 ug (Part 2 Period 2), and MK-5475 240 ug (Part 2 Period 3).
- MK-5475 120 ug/MK-5475 165 ug/Placebo/MK-5475 240 ug/MK-5475 240 ug (Panel A): Participants received inhaled doses as follows: MK-5475 120 ug (Part 1 Period 1), MK-5475 165 ug (Part 1 Period 2), placebo (Part 1 Period 3), MK-5475 240 ug (Part 2 Period 2), and MK-5475 240 ug (Part 2 Period 3).
- Placebo/MK-5475 165 ug/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A): Participant received inhaled doses as follows: placebo (Part 1 Period 1), MK-5475 165 ug (Part 1 Period 2), MK-5475 240 ug (Part 1 Period 3), 240 ug (Part 2 Period 2), and 240 ug (Part 2 Period 3).
- Placebo/MK-5475 165 ug/MK-5475 240 ug (Panel A): Participant received inhaled doses as follows: placebo (Part 1 Period 1), MK-5475 165 ug (Part 1 Period 2), and 240 ug (Part 1 Period 3).
- MK-5475 300 ug/ MK-5475 165 ug/ MK-5475 165 ug (Panel B): Participant received inhaled doses as follows: MK-5475 300 ug (Part 2 Period 1), MK-5475 165 ug (Part 2 Period 2), and 165 ug (Part 2 Period 3).
- MK-5475 300 ug/ MK-5475 360 ug/ MK-5475 360 ug (Panels B+C): Participants received inhaled doses as follows: MK-5475 300 ug (Part 2 Period 1), MK-5475 360 ug (Part 2 Period 2), and 360 ug (Part 2 Period 3).
- MK-5475 300 ug/ MK-5475 120 ug/ MK-5475 120 ug (Panel C): Participants received inhaled doses as follows: MK-5475 300 ug (Part 2 Period 1), MK-5475 120 ug (Part 2 Period 2), and 120 ug (Part 2 Period 3).
- MK-5475 480 ug/ MK-5475 120 ug/ MK-5475 120 ug (Panel D): Participants received inhaled doses as follows: MK-5475 480 ug (Part 2 Period 1), MK-5475 120 ug (Part 2 Period 2), and 120 ug (Part 2 Period 3).
- MK-5475 480 ug/ MK-5475 120 ug (Panel D): Participant received inhaled doses as follows: MK-5475 480 ug (Part 2 Period 1) and MK-5475 120 ug (Part 2 Period 2).
Period: Overall Study
Arm/Group | MK-5475 120 ug/MK-5475 165 ug/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A) | MK-5475 120 ug/Placebo/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A) | MK-5475 120 ug/MK-5475 165 ug/Placebo/MK-5475 240 ug/MK-5475 240 ug (Panel A) | Placebo/MK-5475 165 ug/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A) | Placebo/MK-5475 165 ug/MK-5475 240 ug (Panel A) | MK-5475 300 ug/ MK-5475 165 ug/ MK-5475 165 ug (Panel B) | MK-5475 300 ug/ MK-5475 360 ug/ MK-5475 360 ug (Panels B+C) | MK-5475 300 ug/ MK-5475 120 ug/ MK-5475 120 ug (Panel C) | MK-5475 480 ug/ MK-5475 120 ug/ MK-5475 120 ug (Panel D) | MK-5475 480 ug/ MK-5475 120 ug (Panel D)
Started | 2 | 2 | 2 | 1 | 1 | 1 | 8 | 4 | 3 | 1
Completed | 2 | 2 | 2 | 1 | 1 (Participant did not receive MK-5475 240 ug in Part 2 as planned.) | 1 (Participant received 165 ug in Part 2 Periods 2 and 3, instead of planned 360 ug.) | 8 | 4 (Participants received 120 ug in Part 2 Periods 2 and 3, instead of planned 360 ug.) | 3 | 1 (Participant did not receive 120 ug in Part 2 Period 3 as planned.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-5475 120 ug/MK-5475 165 ug/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A) | MK-5475 120 ug/Placebo/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A) | MK-5475 120 ug/MK-5475 165 ug/Placebo/MK-5475 240 ug/MK-5475 240 ug (Panel A) | Placebo/MK-5475 165 ug/MK-5475 240 ug/MK-5475 240 ug/MK-5475 240 ug (Panel A) | Placebo/MK-5475 165 ug/MK-5475 240 ug (Panel A) | MK-5475 300 ug/ MK-5475 165 ug/ MK-5475 165 ug (Panel B) | MK-5475 300 ug/ MK-5475 360 ug/ MK-5475 360 ug (Panels B+C) | MK-5475 300 ug/ MK-5475 120 ug/ MK-5475 120 ug (Panel C) | MK-5475 480 ug/ MK-5475 120 ug/ MK-5475 120 ug (Panel D) | MK-5475 480 ug/ MK-5475 120 ug (Panel D) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 1 | 1 | 8 | 4 | 3 | 1 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (1.4) | 51.0 (4.2) | 61.0 (4.2) | 61.0 (NA) — NA = Standard Deviation not reported when n<2. | 61.0 (NA) — NA = Standard Deviation not reported when n<2. | 52.0 (NA) — NA = Standard Deviation not reported when n<2. | 48.6 (14.4) | 61.3 (2.2) | 62.7 (5.9) | 69.0 (NA) — NA = Standard Deviation not reported when n<2. | 55.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 0 | 1 | 0 | 6 | 3 | 2 | 1 | 18
  Male | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 1 | 1 | 1 | 8 | 4 | 3 | 1 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 1 | 1 | 1 | 8 | 4 | 3 | 1 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least 1 Adverse Event (AE): All Parts
Description: An AE was defined as any untoward medical occurrence in a participant which may not necessarily have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease that was temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The number of participants who experienced at least 1 AE was reported by dose separately for Part 1 plus Part 2 Period 1, for the RHC Period, and for the FRI Period.
Time Frame: Up to ~14 days after last dose of treatment period (Up to ~32 weeks total)
Population: All participants who received ≥1 dose of investigational treatment were analyzed according to treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- MK-5475 120 ug: Part 1 (Panel A): Participants received MK-5475 120 ug during Part 1.
- MK-5475 165 ug: Part 1 (Panel A): Participants received MK-5475 165 ug during Part 1.
- MK-5475 240 ug: Part 1 (Panel A): Participants received MK-5475 240 ug during Part 1.
- MK-5475 300 ug: Part 2 Period 1 (Panels B+C): Participants received MK-5475 300 ug during Part 2 Period 1.
- MK-5475 480 ug: Part 2 Period 1 (Panel D): Participants received MK-5475 480 ug during Part 2 Period 1.
- Placebo: Part 1: Participants received placebo during Part 1.
- MK-5475 120 ug: RHC (Panel D): Participants received MK-5475 120 ug during the RHC Period.
- MK-5475 165 ug: RHC (Panel B): Participant received MK-5475 165 ug during the RHC Period.
- MK-5475 240 ug: RHC (Panel A): Participants received MK-5475 240 ug during the RHC Period.
- MK-5475 360 ug: RHC (Panels B+C): Participants received MK-5475 360 ug during the RHC Period.
- MK-5475 120 ug: FRI (Panels C+D): Participants received MK-5475 120 ug during the FRI Period.
- MK-5475 165 ug: FRI (Panel B): Participant received MK-5475 165 ug during the FRI Period.
- MK-5475 240 ug: FRI (Panel A): Participants received MK-5475 240 ug during the FRI Period.
- MK-5475 360 ug: FRI (Panels B+C): Participants received MK-5475 360 ug during the FRI Period.
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panels B+C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panels B+C) | MK-5475 120 ug: FRI (Panels C+D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panels B+C)
Number analyzed (Participants) | 6 | 6 | 6 | 13 | 4 | 6 | 7 | 1 | 7 | 8 | 8 | 1 | 7 | 8
Participants | 2 | 1 | 3 | 5 | 2 | 4 | 5 | 1 | 6 | 4 | 1 | 0 | 0 | 4

2. Primary Outcome: Number of Participants Who Discontinued From the Study Due to an AE: All Parts
Description: An AE was defined as any untoward medical occurrence in a participant which may not necessarily have a causal relationship with the treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease that was temporally associated with use of a medicinal product, regardless of whether or not it was considered related to the medicinal product. The number of participants who discontinued from the study due to an AE was reported by dose separately for Part 1 plus Part 2 Period 1, for the RHC Period, and for the FRI Period.
Time Frame: Up to ~14 days after last dose of treatment period (Up to ~32 weeks total)
Population: All participants who received ≥1 dose of investigational treatment were analyzed according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panels B+C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panels B+C) | MK-5475 120 ug: FRI (Panels C+D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panels B+C)
Number analyzed (Participants) | 6 | 6 | 6 | 13 | 4 | 6 | 7 | 1 | 7 | 8 | 8 | 1 | 7 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage Change From Baseline in Minimum Pulmonary Vascular Resistance (PVR): Part 2 Right Heart Catheterization (RHC) Period
Description: For each participant in the RHC Period, the percentage change from baseline for the minimum post-dose PVR value over the duration of the RHC procedure was calculated. The average of pre-dose measurements was set as the baseline. Mean (SD) percent change from baseline in PVR minimum were calculated and reported for each dose group that underwent RHC in Part 2. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and up to 4.5 hours post-dose
Population: All participants who received ≥1 dose of MK-5475, who complied with the protocol without major protocol deviations, and who underwent the RHC procedure and had available data were analyzed according to treatment received.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panels B+C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panels B+C) | MK-5475 120 ug: FRI (Panels C+D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panels B+C)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 7 | 8 | 0 | 0 | 0 | 0
Percentage change |  |  |  |  |  |  | -20.77 (13.88) | 13.01 (NA) — NA = Standard Deviation not reported when n<2. | -29.46 (13.72) | -29.25 (17.58) |  |  |  |

4. Secondary Outcome: Change From Baseline in Heart Rate (HR) at 0.5 Hours Post-dose: Part 2 RHC Period
Description: HR was assessed at pre-dose in the RHC Period (baseline) and at 0.5 hours post-dose. Baseline HR and change from baseline in HR was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in HR. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 0.5 hours post-dose
Population: All participants who received ≥1 dose of MK-5475, underwent the RHC procedure, and had available data were analyzed. One Panel B participant received 165 ug instead of 360 ug but was included in the 360 ug RHC group. Four Panel C participants were dose-reduced from 360 to 120 ug but were included in the 360 ug RHC group.
Measure: Mean (Standard Error); unit: beats/minute
Groups:
- MK-5475 120 ug: Part 1: Participants received MK-5475 120 ug during Part 1.
- MK-5475 165 ug: Part 1: Participants received MK-5475 165 ug during Part 1.
- MK-5475 240 ug: Part 1: Participants received MK-5475 240 ug during Part 1.
- MK-5475 300 ug: Part 2 Period 1: Participants received MK-5475 300 ug during Part 2 Period 1.
- MK-5475 480 ug: Part 2 Period 1: Participants received MK-5475 480 ug during Part 2 Period 1.
- MK-5475 360 ug: RHC (Panel B): Participants in Panel B received MK-5475 360 ug during the RHC Period.
- MK-5475 360 ug: RHC (Panel C): Participants in Panel C received MK-5475 360 ug during the RHC Period.
- MK-5475 120 ug: FRI: Participants received MK-5475 120 ug during the FRI Period.
- MK-5475 240 ug: FRI: Participants received MK-5475 240 ug during the FRI Period.
- MK-5475 360 ug: FRI: Participants received MK-5475 360 ug during the FRI Period.
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
beats/minute
  Baseline HR |  |  |  |  |  |  | 74.75 (9.78) |  | 62.57 (6.23) | 68.75 (2.36) | 69.06 (4.29) |  |  |  |
  Change from Baseline in HR: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 6 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in HR |  |  |  |  |  |  | 3.56 (7.60) |  | 1.83 (1.56) | 4.92 (3.03) | -2.76 (1.60) |  |  |  |

5. Secondary Outcome: Change From Baseline in Heart Rate (HR) at 4.5 Hours Post-dose: Part 2 RHC Period
Description: HR was assessed at pre-dose in the RHC Period (baseline) and at 4.5 hours post-dose. Baseline HR and change from baseline in HR was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in HR. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 4.5 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Error); unit: beats/minute
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
beats/minute
  Baseline HR |  |  |  |  |  |  | 74.75 (9.78) |  | 62.57 (6.23) | 68.75 (2.36) | 69.06 (4.29) |  |  |  |
  Change from Baseline in HR: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 5 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in HR |  |  |  |  |  |  | -0.56 (4.55) |  | 3.20 (3.51) | 7.17 (1.55) | -0.98 (2.01) |  |  |  |

6. Secondary Outcome: Change From Baseline in Heart Rate (HR) at 24 Hours Post-dose: Part 2 RHC Period
Description: HR was assessed at pre-dose in the RHC Period (baseline) and at 24 hours post-dose. Baseline HR and change from baseline in HR was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in HR. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Error); unit: beats/minute
Groups:
- MK-5475 165 ug: RHC (Panel B): Participants received MK-5475 165 ug during the RHC Period.
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
beats/minute
  Baseline HR |  |  |  |  |  |  | 74.75 (9.78) |  | 62.57 (6.23) | 68.75 (2.36) | 69.06 (4.29) |  |  |  |
  Change from Baseline in HR: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in HR |  |  |  |  |  |  | 1.78 (7.35) |  | 7.43 (3.32) | 2.42 (3.10) | -0.72 (2.53) |  |  |  |

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at 0.5 Hours Post-dose: Part 2 RHC Period
Description: SBP was assessed at pre-dose in the RHC Period (baseline) and at 0.5 hours post-dose. Baseline SBP and change from baseline in SBP was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in SBP. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 0.5 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
Millimeters of mercury (mmHg)
  Baseline SBP |  |  |  |  |  |  | 123.25 (9.80) |  | 132.86 (3.79) | 128.50 (9.65) | 119.11 (4.72) |  |  |  |
  Change from Baseline in SBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 6 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in SBP |  |  |  |  |  |  | 25.33 (2.52) |  | 2.67 (3.70) | -1.17 (3.46) | 5.30 (2.36) |  |  |  |

8. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at 4.5 Hours Post-dose: Part 2 RHC Period
Description: SBP was assessed at pre-dose in the RHC Period (baseline) and at 4.5 hours post-dose. Baseline SBP and change from baseline in SBP was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in SBP. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 4.5 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
Millimeters of mercury (mmHg)
  Baseline SBP |  |  |  |  |  |  | 123.25 (9.80) |  | 132.86 (3.79) | 128.50 (9.65) | 119.11 (4.72) |  |  |  |
  Change from Baseline in SBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 5 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in SBP |  |  |  |  |  |  | 10.67 (0.38) |  | 4.93 (5.65) | 7.50 (1.55) | 11.96 (6.31) |  |  |  |

9. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at 24 Hours Post-dose: Part 2 RHC Period
Description: SBP was assessed at pre-dose in the RHC Period (baseline) and at 24 hours post-dose. Baseline SBP and change from baseline in SBP was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in SBP. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
Millimeters of mercury (mmHg)
  Baseline SBP |  |  |  |  |  |  | 123.25 (9.80) |  | 132.86 (3.79) | 128.50 (9.65) | 119.11 (4.72) |  |  |  |
  Change from Baseline in SBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in SBP |  |  |  |  |  |  | 6.22 (5.28) |  | -5.95 (5.78) | 2.25 (7.62) | 0.74 (3.44) |  |  |  |

10. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at 0.5 Hours Post-dose: Part 2 RHC Period
Description: DBP was assessed at pre-dose in the RHC Period (baseline) and at 0.5 hours post-dose. Baseline DBP and change from baseline in DBP was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in DBP. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 0.5 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
Millimeters of mercury (mmHg)
  Baseline DBP |  |  |  |  |  |  | 69.75 (4.03) |  | 72.43 (2.25) | 77.00 (4.95) | 70.78 (3.52) |  |  |  |
  Change from Baseline in DBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 6 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in DBP |  |  |  |  |  |  | 4.00 (4.60) |  | 0.94 (1.68) | 0.75 (3.48) | 1.30 (1.75) |  |  |  |

11. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at 4.5 Hours Post-dose: Part 2 RHC Period
Description: DBP was assessed at pre-dose in the RHC Period (baseline) and at 4.5 hours post-dose. Baseline DBP and change from baseline in DBP was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in DBP. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 4.5 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
Millimeters of mercury (mmHg)
  Baseline DBP |  |  |  |  |  |  | 69.75 (4.03) |  | 72.43 (2.25) | 77.00 (4.95) | 70.78 (3.52) |  |  |  |
  Change from Baseline in DBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 5 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in DBP |  |  |  |  |  |  | -0.22 (4.87) |  | 1.07 (2.34) | 3.58 (2.73) | 4.00 (4.28) |  |  |  |

12. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at 24 Hours Post-dose: Part 2 RHC Period
Description: DBP was assessed at pre-dose in the RHC Period (baseline) and at 24 hours post-dose. Baseline DBP and change from baseline in DBP was reported for each panel/dose group that underwent RHC in Part 2, according to treatment planned. Negative values indicate decreases from baseline in DBP. Per protocol, this outcome measure was only assessed during the Part 2 RHC Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of RHC Period (up to 185 days) and 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | MK-5475 120 ug: Part 1 | MK-5475 165 ug: Part 1 | MK-5475 240 ug: Part 1 | MK-5475 300 ug: Part 2 Period 1 | MK-5475 480 ug: Part 2 Period 1 | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI | MK-5475 360 ug: FRI
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
Millimeters of mercury (mmHg)
  Baseline SBP |  |  |  |  |  |  | 69.75 (4.03) |  | 72.43 (2.25) | 77.00 (4.95) | 70.78 (3.52) |  |  |  |
  Change from Baseline in SBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 7 | 4 | 9 | 0 | 0 | 0 | 0
  Change from Baseline in SBP |  |  |  |  |  |  | -1.44 (0.89) |  | -2.76 (3.22) | 2.42 (3.15) | -1.74 (2.89) |  |  |  |

13. Secondary Outcome: Area Under the Concentration-Time Curve From Hour 0 to Infinity (AUC0-inf) of MK-5475: All Parts
Description: Blood samples were taken at predose and at specified time points postdose to determine the AUC0-inf of MK-5475. AUC0-inf was defined as the area under the concentration-time curve of MK-5475 from time zero to infinity. MK-5475 AUC0-inf was reported by panel/dose group. Per protocol, percent geometric coefficient of variation (%GCV) values were not reported for groups with n<2 participants.
Time Frame: Part 1 and Part 2 Period 1: Predose and 0.1, 0.25, 0.5, 1, 2, 3, 4, 8, and 24 hours post-dose; RHC Period: predose and 0.25, 0.5, 1, 2, 3, 4, and 4.5 hours; FRI Period: predose and 1, 3, 8, and 24 hours postdose (Panel D also 0.25, 0.5, 2, 4 hours)
Population: All participants who received at least one dose of MK-5475, who complied with the protocol without major protocol deviations, and who had available data for AUC0-inf were analyzed. Per protocol, data from participants receiving placebo were not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Groups:
- MK-5475 120 ug: Part 1 (Panel A): Participants in Panel A received MK-5475 120 ug during Part 1.
- MK-5475 165 ug: Part 1 (Panel A): Participants in Panel A received MK-5475 165 ug during Part 1.
- MK-5475 240 ug: Part 1 (Panel A): Participants in Panel A received MK-5475 240 ug during Part 1.
- MK-5475 300 ug: Part 2 Period 1 (Panel B): Participants in Panel B received MK-5475 300 ug during Part 2 Period 1.
- MK-5475 300 ug: Part 2 Period 1 (Panel C): Participants in Panel C received MK-5475 300 ug during Part 2 Period 1.
- MK-5475 480 ug: Part 2 Period 1 (Panel D): Participants in Panel D received MK-5475 480 ug during Part 2 Period 1.
- MK-5475 120 ug: RHC (Panel C): Participants in Panel C received MK-5475 120 ug during the RHC Period.
- MK-5475 120 ug: RHC (Panel D): Participants in Panel D received MK-5475 120 ug during the RHC Period.
- MK-5475 165 ug: RHC (Panel B): Participant in Panel B received MK-5475 165 ug during the RHC Period.
- MK-5475 240 ug: RHC (Panel A): Participants in Panel A received MK-5475 240 ug during the RHC Period.
- MK-5475 120 ug: FRI (Panel C): Participants in Panel C received MK-5475 120 ug during the FRI Period.
- MK-5475 120 ug: FRI (Panel D): Participants in Panel D received MK-5475 120 ug during the FRI Period.
- MK-5475 165 ug: FRI (Panel B): Participant in Panel B received MK-5475 165 ug during the FRI Period.
- MK-5475 240 ug: FRI (Panel A): Participants in Panel A received MK-5475 240 ug during the FRI Period.
- MK-5475 360 ug: FRI (Panel B): Participants in Panel B received MK-5475 360 ug during the FRI Period.
- MK-5475 360 ug: FRI (Panel C): Participants in Panel C received MK-5475 360 ug during the FRI Period.
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panel B) | MK-5475 300 ug: Part 2 Period 1 (Panel C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel C) | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI (Panel C) | MK-5475 120 ug: FRI (Panel D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panel B) | MK-5475 360 ug: FRI (Panel C)
Number analyzed (Participants) | 2 | 5 | 6 | 4 | 9 | 4 | 0 | 4 | 3 | 0 | 6 | 3 | 5 | 3 | 4 | 1 | 0 | 0 | 4
nM*hr | 1.00 (45.5) | 0.721 (103.6) | 1.25 (59.7) | 2.15 (106.3) | 1.66 (66.8) | 4.59 (20.9) |  | 1.03 (20.0) | 1.05 (28.9) |  | 1.03 (59.7) | 1.46 (63.2) | 3.46 (67.3) | 0.748 (43.9) | 0.978 (18.3) | 4.26 (NA) — NA = %GCV values were not reported when n<2 |  |  | 4.10 (37.6)

14. Secondary Outcome: Area Under the Concentration-Time Curve From Hour 0 to 24 Hours (AUC0-24hr) of MK-5475: All Parts
Description: Blood samples were taken at predose and at specified time points postdose to determine the AUC0-24hr of MK-5475. AUC0-24hr was defined as the area under the concentration-time curve of MK-5475 from time zero to 24 hours. MK-5475 AUC0-24hr was reported by panel/dose group. For RHC panel/dose groups where sampling was only done up to 4.5 hours, the AUC0-24hr geometric mean represents an extrapolated AUC0-24hr value. Per protocol, %GCV values were not reported for groups with n<2 participants.
Time Frame: as for outcome 13
Population: All participants who received at least one dose of MK-5475, who complied with the protocol without major protocol deviations, and who had available data for AUC0-24hr were analyzed. Per protocol, data from participants receiving placebo were not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panel B) | MK-5475 300 ug: Part 2 Period 1 (Panel C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel C) | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI (Panel C) | MK-5475 120 ug: FRI (Panel D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panel B) | MK-5475 360 ug: FRI (Panel C)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 9 | 4 | 0 | 4 | 4 | 1 | 7 | 3 | 5 | 4 | 4 | 1 | 7 | 3 | 5
nM*hr | 0.259 (288.2) | 0.613 (136.0) | 1.42 (59.9) | 2.35 (96.2) | 1.82 (63.2) | 4.53 (21.0) |  | 1.02 (18.5) | 1.05 (28.9) | NA (NA) — NA = Not calculated due to insufficient samples on the terminal phase to estimate lambda z | 1.04 (59.0) | 1.45 (61.7) | 3.48 (68.3) | 0.747 (43.5) | 1.13 (18.4) | 4.19 (NA) — NA = %GCV values were not reported when n<2 | 1.71 (43.3) | 1.21 (80.1) | 3.82 (35.3)

15. Secondary Outcome: Maximum Concentration (Cmax) of MK-5475: All Parts
Description: Blood samples were taken at predose and at specified time points postdose to determine the Cmax of MK-5475. Cmax was defined as the maximum concentration of MK-5475 reached. MK-5475 Cmax was reported by panel/dose group. Per protocol, %GCV values were not reported for groups with n<2 participants.
Time Frame: as for outcome 13
Population: All participants who received at least one dose of MK-5475, who complied with the protocol without major protocol deviations, and who had available data for Cmax were analyzed. Per protocol, data from participants receiving placebo were not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panel B) | MK-5475 300 ug: Part 2 Period 1 (Panel C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel C) | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI (Panel C) | MK-5475 120 ug: FRI (Panel D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panel B) | MK-5475 360 ug: FRI (Panel C)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 9 | 4 | 0 | 4 | 4 | 1 | 7 | 3 | 5 | 4 | 4 | 1 | 7 | 3 | 5
nM | 0.0722 (153.3) | 0.139 (117.9) | 0.297 (60.8) | 0.543 (73.9) | 0.409 (66.0) | 0.981 (22.9) |  | 0.218 (4.7) | 0.161 (76.5) | 0.312 (NA) — NA = %GCV values were not reported when n<2 | 0.202 (59.7) | 0.307 (21.7) | 0.960 (67.9) | 0.228 (36.8) | 0.245 (21.7) | 0.601 (NA) — NA = %GCV values were not reported when n<2 | 0.341 (40.1) | 0.301 (69.8) | 0.915 (56.5)

16. Secondary Outcome: Concentration of MK-5475 at 24 Hours Postdose (C24): All Parts
Description: Blood samples were taken at predose and at specified time points postdose to determine the C24 of MK-5475. C24 was defined as the concentration of MK-5475 reached at 24 hours. MK-5475 Cmax was reported by panel/dose group. Per protocol, %GCV values were not reported for groups with n<2 participants.
Time Frame: 24 hours postdose
Population: All participants who received at least one dose of MK-5475, who complied with the protocol without major protocol deviations, and who had available data for C24 were analyzed. Per protocol, data from participants receiving placebo were not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panel B) | MK-5475 300 ug: Part 2 Period 1 (Panel C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel C) | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI (Panel C) | MK-5475 120 ug: FRI (Panel D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panel B) | MK-5475 360 ug: FRI (Panel C)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 9 | 4 | 0 | 4 | 4 | 1 | 7 | 3 | 5 | 4 | 4 | 1 | 7 | 3 | 5
nM | NA (NA) — NA= no participant had detectable C24 | NA (NA) — NA= no participant had detectable C24 | NA (NA) — NA= no participant had detectable C24 | NA (NA) — NA= no participant had detectable C24 | NA (NA) — NA= no participant had detectable C24 | 0.0113 (25.0) |  | NA (NA) — NA = C24 could not be calculated since PK samples were only collected up to 4.5 hours in the RHC Period | NA (NA) — NA = C24 could not be calculated since PK samples were only collected up to 4.5 hours in the RHC Period | NA (NA) — NA = C24 could not be calculated since PK samples were only collected up to 4.5 hours in the RHC Period | NA (NA) — NA = C24 could not be calculated since PK samples were only collected up to 4.5 hours in the RHC Period | NA (NA) — NA = C24 could not be calculated since PK samples were only collected up to 4.5 hours in the RHC Period | NA (NA) — NA = C24 could not be calculated since PK samples were only collected up to 4.5 hours in the RHC Period | NA (NA) — NA= no participant had detectable C24 | NA (NA) — NA= no participant had detectable C24 | 0.0128 (NA) — NA = %GCV values were not reported when n<2 | NA (NA) — NA = C24 could not be calculated due to an insufficient number of participants with detectable C24 to calculate geometric mean (%GCV) | NA (NA) — NA= no participant had detectable C24 | NA (NA) — NA = C24 could not be calculated due to an insufficient number of participants with detectable C24 to calculate geometric mean (%GCV)

17. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-5475: All Parts
Description: Blood samples were taken at predose and at specified time points postdose to determine the Tmax of MK-5475. Tmax was defined as the time to maximum concentration of MK-5475. MK-5475 Tmax was reported by panel/dose group.
Time Frame: as for outcome 13
Population: All participants who received at least one dose of MK-5475, who complied with the protocol without major protocol deviations, and who had available data for Tmax were analyzed. Per protocol, data from participants receiving placebo were not included in the analysis.
Measure: Median (Full Range); unit: Hour
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panel B) | MK-5475 300 ug: Part 2 Period 1 (Panel C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel C) | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI (Panel C) | MK-5475 120 ug: FRI (Panel D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panel B) | MK-5475 360 ug: FRI (Panel C)
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 9 | 4 | 0 | 4 | 4 | 1 | 7 | 3 | 5 | 4 | 4 | 1 | 7 | 3 | 5
Hour | 2.00 [2.00 to 2.00] | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 2.00] | 1.50 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00] |  | 1.00 [0.50 to 1.00] | 1.00 [0.00 to 1.00] | 3.00 [3.00 to 3.00] | 2.00 [1.00 to 3.00] | 1.00 [1.00 to 1.00] | 1.00 [0.50 to 1.00] | 1.00 [1.00 to 3.00] | 1.50 [1.00 to 2.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 1.00]

18. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MK-5475: All Parts
Description: Blood samples were taken at predose and at specified time points postdose to determine the t½ of MK-5475. t½ was defined as the time required to divide the MK-5475 plasma concentration by two after reaching pseudo-equilibrium, following a single dose of MK-5475. MK-5475 t½ was reported by panel/dose group.
Time Frame: as for outcome 13
Population: All participants who received at least one dose of MK-5475, who complied with the protocol without major protocol deviations, and who had available data for t½ were analyzed. Per protocol, data from participants receiving placebo were not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panel B) | MK-5475 300 ug: Part 2 Period 1 (Panel C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel C) | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panel B) | MK-5475 360 ug: RHC (Panel C) | MK-5475 120 ug: FRI (Panel C) | MK-5475 120 ug: FRI (Panel D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panel B) | MK-5475 360 ug: FRI (Panel C)
Number analyzed (Participants) | 2 | 5 | 6 | 4 | 9 | 4 | 0 | 4 | 3 | 0 | 6 | 3 | 5 | 3 | 4 | 1 | 0 | 0 | 4
Hour | 1.73 (11.4) | 1.76 (10.9) | 1.87 (13.5) | 2.12 (37.2) | 2.18 (37.9) | 3.67 (6.6) |  | 2.82 (10.5) | 2.32 (21.0) |  | 2.35 (9.2) | 3.13 (45.5) | 2.05 (11.6) | 2.45 (24.6) | 2.19 (8.1) | 3.89 (NA) — NA = %GCV values were not reported when n<2 |  |  | 3.92 (7.9)

19. Secondary Outcome: Percentage Change From Baseline in Pulmonary Blood Volume (PBV) Over Time: Part 2 Functional Respiratory Imaging (FRI) Period
Description: Participants underwent a series of computed tomography (CT) scans with an intravenous (IV) iodinated contrast agent to facilitate assessment of PBV at baseline and at several times points after MK-5475 dosing. Percentage change from baseline (CFB) in PBV was calculated and reported for each dose group that underwent FRI in Part 2. As pre-specified, central tendency for PBV percentage CFB was provided as numerical values rounded to whole numbers. Per protocol, this outcome measure was only assessed during the Part 2 FRI Period for each panel and was not assessed during Part 1.
Time Frame: Baseline: Pre-dose on Day 1 of FRI Period (up to 227 days) and 1, 3, 8, and 24 hours post-dose
Population: All participants who received MK-5475 at 120, 240 or 360 ug during the FRI period and underwent CT scans with IV contrast agent at all time points were included in the analysis.
Measure: Number; unit: Percentage change
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panels B+C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panels B+C) | MK-5475 120 ug: FRI (Panels C+D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panels B+C)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 6 | 7
Percentage change
  CFB at 1 hour |  |  |  |  |  |  |  |  |  |  | -2 |  | 2 | 3
  CFB at 3 hours |  |  |  |  |  |  |  |  |  |  | 2 |  | 2 | 9
  CFB at 8 hours |  |  |  |  |  |  |  |  |  |  | 3 |  | 11 | 9
  CFB at 24 hours |  |  |  |  |  |  |  |  |  |  | -2 |  | 3 | 6

ADVERSE EVENTS:
Time Frame: Up to ~14 days after last dose of treatment period (Up to ~32 weeks total)
Description: All-Cause Mortality table includes all randomized participants. Serious and Other adverse events (AEs) tables include all randomized participants who received at least 1 dose of study drug.
Arm/Group | MK-5475 120 ug: Part 1 (Panel A) | MK-5475 165 ug: Part 1 (Panel A) | MK-5475 240 ug: Part 1 (Panel A) | MK-5475 300 ug: Part 2 Period 1 (Panels B+C) | MK-5475 480 ug: Part 2 Period 1 (Panel D) | Placebo: Part 1 | MK-5475 120 ug: RHC (Panel D) | MK-5475 165 ug: RHC (Panel B) | MK-5475 240 ug: RHC (Panel A) | MK-5475 360 ug: RHC (Panels B+C) | MK-5475 120 ug: FRI (Panels C+D) | MK-5475 165 ug: FRI (Panel B) | MK-5475 240 ug: FRI (Panel A) | MK-5475 360 ug: FRI (Panels B+C)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/13 | 0/4 | 0/6 | 0/7 | 0/1 | 0/7 | 0/8 | 0/8 | 0/1 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/13 | 0/4 | 0/6 | 0/7 | 0/1 | 0/7 | 0/8 | 0/8 | 0/1 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 3/6 | 5/13 | 2/4 | 4/6 | 5/7 | 1/1 | 6/7 | 4/8 | 1/8 | 0/1 | 0/7 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5475 120 ug: Part 1 (Panel A) (N=6) | MK-5475 165 ug: Part 1 (Panel A) (N=6) | MK-5475 240 ug: Part 1 (Panel A) (N=6) | MK-5475 300 ug: Part 2 Period 1 (Panels B+C) (N=13) | MK-5475 480 ug: Part 2 Period 1 (Panel D) (N=4) | Placebo: Part 1 (N=6) | MK-5475 120 ug: RHC (Panel D) (N=7) | MK-5475 165 ug: RHC (Panel B) (N=1) | MK-5475 240 ug: RHC (Panel A) (N=7) | MK-5475 360 ug: RHC (Panels B+C) (N=8) | MK-5475 120 ug: FRI (Panels C+D) (N=8) | MK-5475 165 ug: FRI (Panel B) (N=1) | MK-5475 240 ug: FRI (Panel A) (N=7) | MK-5475 360 ug: FRI (Panels B+C) (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign enlargement of the subarachnoid spaces (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT03744637/Prot_SAP_000.pdf